CLINICAL TRIAL: NCT04240795
Title: The Effects of Hydrogels Differing in Their Lubricity on Appetite Control, Satiety, Subsequent Food Intake and Salivary Biomarkers
Brief Title: Effect of Lubricity of Food Gels on Satiation and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Anwesha Sarkar, Associate Professor, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LUBSAT (18-049)
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Appetitive Behavior
Keywords: Food Structure; Gel; Satiety; Appetite; Food intake; Salivary biomarkers; Mucin; Amylase; Hunger; Fullness
MeSH Terms: conditions — Appetitive Behavior; Medullary cystic kidney disease 1 | interventions — Water

STUDY DESIGN:
Intervention Model Description: Tightly controlled cross-over study design with three arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low lubricity (LL) hydrogels containing fibre-based beads (Experimental): Participants are given a preload of 30 g of low lubricity hydrogels (alginate beads in kappa-carrageenan hydrogels) after 2.5 hours after a standardized breakfast. After 30 minutes of the preload, participants are given ad libitum lunch. They are asked to eat "as much or as little as they want, until they feel comfortably full".
  Interventions: Dietary Supplement: Low lubricity (LL) hydrogels containing fibre-based beads
- High lubricity (HL) hydrogels containing no fibre-based beads (Active Comparator): Participants are given a preload of 30 g of high lubricity hydrogels (no beads in kappa-carrageenan and alginate mixed hydrogels) after 2.5 hours after a standardized breakfast. After 30 minutes of the preload, participants are given ad libitum lunch. They are asked to eat "as much or as little as they want, until they feel comfortably full".
  Interventions: Dietary Supplement: Low lubricity (LL) hydrogels containing fibre-based beads
- Water (Placebo Comparator): The water containing the same watermelon flavor, color and sweetness was given as control to match the gels. Participants receive the same amount of water like hydrogels - 30 g after 2.5 hours after a standardized breakfast. After 30 minutes of the preload, participants are given ad libitum lunch. They are asked to eat "as much or as little as they want, until they feel comfortably full".
  Interventions: Dietary Supplement: Low lubricity (LL) hydrogels containing fibre-based beads

INTERVENTIONS:
Dietary Supplement: Low lubricity (LL) hydrogels containing fibre-based beads — The preload is made from kappa-carrageenan and alginate beads of 450 μm size. It contains no additional macronutrient but has food-grade watermelon flavor, color, and non-nutritive sweetener.
  Other Names: High lubricity (HL) hydrogels containing no fibre-based beads; Water

SUMMARY:
The main aim of the study is to elucidate the influence of fibre-based hydrogels differing in their mechanical properties (characterized both instrumentally and sensorially) in terms of low/ high lubricity on satiety, satiation and salivary biomarkers.

DETAILED DESCRIPTION:
An acute, randomized cross-over study that compares two types of fibre-based hydrogels differing in their lubrication properties, resulting in different pastiness and instrumental mechanical properties (lubricity). The gels are prepared using dietary fibres (kappa carrageenan, alginate). Both hydrogels contain added watermelon flavor, food grade color and sweetener. Water acts as a control and has the same flavor, color and sweetness to match the hydrogels.

Participants are asked come to the laboratory on three occasions. Before participating, each participant is screened for eligibility criteria using an online health screening questionnaire and Three Factors Eating Questionnaire. Participants are offered one of the three products (water or either of the two gels), the order of which is randomized and counterbalanced.

Participants are instructed to fast for 11 hours and to restrict from drinking alcohol for 24 hours before each session. In the first session, weight and height are measured. Participants then provide baseline (- 5 minutes) appetite ratings on a 100 mm visual analogue scale (VAS). After that they are given a standardized breakfast (females - 250kcal, males - 350 kcal). Then, participants are asked to rate their appetite on a 100-mm VAS in every 30 minutes for the next 2.5 hours. After that, they are given the preload - either hydrogels differing in their structure complexity or water. After consuming the preload, appetite ratings are recorded by the participants on three time points on 100-mm VAS. Ad libitum food is offered as lunch after 30 minutes after ingesting the preload and the last VAS is taken. Food intake is measured. Saliva is taken three times during each session after breakfast, before and after preload consumption to measure protein, mucin content, amylase activity, and salivary lubricity (tribology).

ELIGIBILITY:
Inclusion Criteria:

* With a normal weight (BMI=18.5 - 24.99 kg/m²)
* Generally healthy

Exclusion Criteria:

* A smoker
* Having oral infections/diseases/problems in chewing and swallowing
* Anyone with a chronic or acute health condition that may affect the ability to sense, eat, digest or absorb food
* Anyone currently using prescribed or non-prescribed medication that may interfere with the ability to sense, eat, digest or absorb food
* Anyone who is pregnant or lactating
* Anyone with a food allergy or intolerance
* Anyone who are on a special diet or are taking protein/fiber supplements
* Anyone who cannot tolerate food gels
* Underweight (BMI <18.5 kg/m²) or overweight (25 - 29.99 kg/m²) or obese (BMI=>29.99 kg/m²)
* Suffer from any blood borne disease e.g. HIV, Hep B

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Baseline level and change in hunger ratings | -5 minutes, 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 160 minutes, 170 minutes, 180 minutes, 190 minutes, 225 minutes
  A questionnaire assessing perceived hunger is completed at specific times points throughout each of the 3.5-hours testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks : "How hungry do you feel right now?" with anchors of "not all" to "extremely." The range is 0 mm (min hunger) and 100 is (max hunger).
Baseline level and change in fullness ratings | -5 minutes, 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 160 minutes, 170 minutes, 180 minutes, 190 minutes, 225 minutes
  A questionnaire assessing perceived fullness is completed at specific time points throughout each of the 3.5-hours testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How full do you feel right now?" with anchors of "not all" to "extremely." The range is 0 mm (min fullness) and 100 is (max fullness).
Baseline level and change in desire to eat ratings | -5 minutes, 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 160 minutes, 170 minutes, 180 minutes, 190 minutes, 225 minutes
  A questionnaire assessing perceived desire to eat is completed at specific time points throughout each of the 3.5-hours testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How strong is your desire to eat right now?" with anchors of "not all" to "extremely." The range is 0 mm (min desire to eat) and 100 is (max desire to eat)
Baseline level and change in prospective food consumption ratings | -5 minutes, 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 160 minutes, 170 minutes, 180 minutes, 190 minutes, 225 minutes
  A questionnaire assessing perceived prospective food consumption is completed at specific time points throughout each of the 3.5-hours testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How much food do you think you could eat right now?" with anchors of "not all" to "extremely." The range is 0 mm (min prospective food consumption) and 100 is (max prospective food consumption).
Baseline level and change in thirst ratings | -5 minutes, 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 160 minutes, 170 minutes, 180 minutes, 190 minutes, 225 minutes
  A questionnaire assessing perceived thirst is completed at specific time points throughout each of the 3.5-hours testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How thirsty do you feel right now?" with anchors of "not all" to "extremely." The range is 0 mm (min thirst) and 100 is (max thirst).
Energy Intake | 20 minutes after the preload
  The participants are provided with an ad libitum lunch of rice and vegetables, strawberry yogurt water. The amount of lunch is provided (in grams) and is weighted prior to consumption and any remains are re-weighted after consumption. Energy consumed will be calculated.
Baseline level and change in salivary properties | 90 minutes, 150 minutes, 170 minutes
  Saliva is collected on three time points on each visit. Salivary protein, amylase, mucin and statherin will be analysed and salivary lubricity will be mesaured

SECONDARY OUTCOMES:
Palatibility of the preloads | Immediately after eating the preload
  The palatability of both the hydrogels and water are assessed through a 100 mm VAS scale. Within the palatability the ratings are taking on following attributes: the texture, flavor and sweetness. The questions asked are: "How much did you like the texture of the product you have just eaten?", "How much did you like the flavor of the product you have just eaten?", How intense was the sweet taste of the product you have just eaten?" with anchors from "not at all" to "extremely".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No